CLINICAL TRIAL: NCT00590746
Title: Bedside Assessment of Fall Risk in Emergency Department Elders
Status: Completed | Type: Observational
Sponsor: Jeffrey Caterino (Other)
Responsible Party: Sponsor-Investigator, Jeffrey Caterino, Assistant Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2007H0239
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Accidental Falls

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the risk for falls among elderly Emergency Department (ED) patients.This study will use 2 tests of balance, the Bertec Balance Screening Test and the "Up and Go" test. These tests measure how steady a person is while standing, walking, and turning 180 degrees. After patients have returned home, they will be contacted at 7 days, 30 days and 6 months to determine if they have sustained a fall during these intervals in order to find out how predictive the balance tests are in determining the risk of future falls.

DETAILED DESCRIPTION:
Falls are one of the most significant health risks to older Americans. In the U.S., 30-60% of community dwelling elders will fall each year.Studies have found rates of serious injury among elders who fall to range from 5-24%. Five percent of those who fall are hospitalized. Among elders, falls cause 2/3 of the deaths due to unintentional injury, the 6th leading cause of death in this age group. Additional major morbidity due to falls includes loss of independence as well as anxiety due to fear of falling. This results in limitation of function and often in a requirement for long-term care. Up to 40% of nursing home admissions are due to falls or fear of falling. Expenditures for fall-related injuries account for 6% of all medical expenditures in geriatric patients. Several interventions have been proven effective to reduce rates of fall. Implementation of these interventions requires physician appreciation of the risk for falls in individual patients. The emergency department (ED) may provide a location to identify patients at increased risk of falling. Unfortunately, successful ED based studies to identify and intervene on at-risk elders have been rare and not widely reproducible. The results of these previous ED studies demonstrate that a rapid, efficient, measurable assessment of balance is required if emergency physicians are to regularly consider such factors in their care plans and disposition decisions. Development of a single, simple screening test to identify ED elders at who fall may improve falls screening in the ED and prevent unnecessary morbidity and mortality by facilitating early identification and intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age > 59 years
* Discharge from Emergency Department
* Self-reported weight < 300 pounds
* Patient resides in the community or a personal care home
* Patients must also confirm that they are able to walk 30 feet without help of another person.They may do this with use of an assistive device.

Exclusion Criteria:

* Age <60 years
* Subject is incarcerated
* Non-English speaking
* Lack of ability of patient to give consent or complete the study tasks
* Patient resides in a nursing home or rehabilitation facility
* Primary evaluation by the trauma team
* Inability to walk 30 feet without assistance from another person

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 60 and older who present to the Ohio State University Medical Center Emergency Department
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2007-12; Primary Completion 2008-10 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To determine the accuracy of the timed Timed Up-and-go test in the ED | 1 year
To determine the accuracy of the Bertec BalanceCheck Screener system in the ED. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Caterino, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center Emergency Department, Columbus, Ohio, United States